CLINICAL TRIAL: NCT05400135
Title: Qungasvik (Toolbox): Prevention of Alcohol/Suicide Risk in Alaska Native Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alaska Fairbanks (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01AA023754 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Suicide; Alcohol Use Disorder
Keywords: Alaska Native; Alcohol; Indigenous; Rural; Suicide; Prevention; Multi-level; Small samples; Dynamic wait-listed design; Stepped wedge design; Protective Factors; Reasons for Life
MeSH Terms: conditions — Suicide; Alcoholism

STUDY DESIGN:
Intervention Model Description: The study utilizes a hybrid design with a two group community level four year interrupted time series design with an embedded five group community level dynamic wait-listed design. Youth participants (12-18 years) in each community are assigned to a single treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qungasvik Intervention Group (Experimental): Qungasvik implements intervention modules creating episodes of Yup'ik cultural engagement. In traditional Yup'ik practices prior to formal western schooling, the education and training of young people included introduction to cultural protocols, knowledge, and values while learning skills through participation in daily activities of family and community life such as subsistence, tool-building, and ceremony (Rasmus, Charles, & Mohatt, 2014). The intervention manual provides outlines for 18 modules described as teachings, and conducted at the individual, family, or community level through one or more 1-3 hour sessions. Each module promotes 2-4 of a total of 13 protective factors.
  Interventions: Behavioral: Qungasvik (Tools for Life)

INTERVENTIONS:
Behavioral: Qungasvik (Tools for Life) — The Qungasvik (toolbox) intervention is designed to build protection against alcohol use disorder (AUD) and suicide in Yup'ik Alaska Native youth 12-18 years old. The intervention is a community-driven and culturally-based process that develops and delivers 18-24 prevention activities leading to the two primary prevention variables, Reasons for Life and Reflective Processes about the Consequences of Alcohol Use and secondary prevention variables of multi-level protective factors and social networks.

SUMMARY:
For the past 20+ years the investigators have focused on addressing two interrelated public health issues, alcohol use disorder (AUD) and suicide in Alaska. There is no greater source of health disparity in American Indian and Alaska Native (AI/AN) communities than that involving AUD and suicide, and no greater necessity in addressing this disparity than the development of sustained, trusting, collaborative, and non-exploitive research relationships with those who historically experienced forced acculturation and exploitation. Yup'ik community leaders have made addressing AUD and suicide among their highest priorities. Working with Yup'ik community members, the investigators developed a multilevel (individual, family, peer, and community) intervention that uses a culturally-based AUD and suicide prevention framework. The Qungasvik (kung-az-vik; a Yup'ik word meaning 'toolbox') intervention is a Yup'ik AN approach to prevention organized and implemented utilizing a local indigenous theory of change and process model to build protective factors against AUD and suicide. The purposes of the proposed research are to: (a) validate results obtained from previous smaller intervention studies aimed at reducing the incidence of AUD and suicide in 12-18 year old Yup'ik Alaska Native (AN) youth; and (b) learn more about the relative importance of the individual, family, peer, and community variables that underscore the Qungasvik intervention. This study will: (a) assess the efficacy of the Qungasvik intervention through a two group community level trial using an interrupted time series design with wait-listed control, and (b) examine mechanisms of change in response to intervention. Specific aims (SA) of the project are to: (SA1) test the Qungasvik intervention efficacy through impact on the ultimate outcome variables of reasons for life and reflective processes on alcohol use consequences, and on suicidal ideation and alcohol use; (SA2) examine the mechanisms of change in response to the Qungasvik intervention through (a) self-report outcome measures of protective factors (b) social network assessment and (c) process evaluation; (SA3) test levels of fidelity of the implementation of the intervention with regard to the Yup'ik indigenous theory-driven intervention model outlined in the Qungasvik manual of operations.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native youth 12-21 years

Exclusion Criteria:

* Children under the age of 12

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 542 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Reflective Processes | Baseline, 1-year, 2-year, 3-year, 4-year
  5 items, item separation reliability=.77. This measure is adapted from the adult Yup'ik Protective Factors scale5, and taps a culturally patterned type of awareness (ellangneq) used in thinking over potential negative consequences of alcohol misuse engaged by Alaska Native youth when considering reasons to not drink.
Change in Reasons for Life | Baseline, 1-year, 2-year, 3-year, 4-year
  5 items, =.78. This measure is an extension of constructs tapped in the Brief Reasons for Living Inventory for Adolescents, itself a modification of an adult measure, the Reasons for Living Inventory. RFL assess beliefs and experiences that make life enjoyable, worthwhile, and provide meaning. Items tap cultural/spiritual beliefs, sense of family responsibility, and others' assessment of the young person. The measure provides a positive psychology approach to assessing AN cultural values associated with protection from suicide.
Change in Alcohol Consequences | Baseline, 1-year, 2-year, 3-year, 4-year
  The five-item CoNcise Inventory of Problems for Alaska Native Adolescents (NIP-AN-A), adaptation of the Adult NIP-AN, taps social, intrapersonal, impulse control, interpersonal and kinship loss. We adapted the Alcohol Quantity/Frequency/Binge Episode Measure (Q-F-BE) for use in rural Alaska. It assesses the quantity and frequency of drinking including binge drinking episodes which are defined as a consumption pattern of greater than four drinks on one occasion.
Change in Rollnick's Readiness Ruler | Baseline, 1-year, 2-year, 3-year, 4-year
  An adaptation of the RRR will provide an analog scale assessment of motivation to remain abstinent.

SECONDARY OUTCOMES:
Change in Individual Protective Factors | Baseline, 1-year, 2-year, 3-year, 4-year
  (10 items, alpha=.69). This uses the Mastery-Family and Mastery-Friends subscales from the Multicultural Mastery Scale to measure communal mastery, or efficacy in solving life challenges and control through strategies that focus on joining with other significant figures in the social environment.
Change in Family Protective Factors | Baseline, 1-year, 2-year, 3-year, 4-year
  (19 items, alpha=.69). The Brief Family Relationship Scale includes subscales tapping Cohesion, Expressiveness, and Conflict, and was designed as a culturally appropriate adaptation of the Family Environment Scale relationship dimension.
Change in Community Protective Factors | Baseline, 1-year, 2-year, 3-year, 4-year
  (7 items, alpha=.62). The Youth Community Protective Factors Scale was adapted from the Yup'ik Protective Factors scale5 to measure elements of protective communities for youth. Its subscales tap Support and Opportunities for youth in their community.
Change in Peer Influences | Baseline, 1-year, 2-year, 3-year, 4-year
  (10 items, alpha=.96). Peer Influences was adapted for understandability and relevance to rural AN youth from the American Drug and Alcohol Survey which has been used extensively in research with American Indian youth on peer attitudes that discourage alcohol use.

OTHER OUTCOMES:
Change in Social Relationships | Baseline through end of intervention delivery, an average of 2 years
  This is a measure that examines social network characteristics of supportive relationships with elders, immediate and extended kinship relations, and community adults.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alaska Fairbanks, Fairbanks, Alaska, United States

IPD SHARING:
Plan to Share IPD: No
Pursuant to Title 45 CFR 46, American Indian and Alaska Native Tribes have the authority to make the decisions and set policy in the protection of human subjects involved in research taking place with members of federally-recognized Tribes. All potential participants in the awarded application are members of federally-recognized Tribes, and each partnering Tribal organization, has passed a formal Resolution or equivalent Tribal law that delegates the ruling body's authority to each of their respective research review boards. The Tribal research review boards will issue binding findings about the proposed research study to include data sharing, ownership and management.